CLINICAL TRIAL: NCT05485688
Title: Impact of Intermittent Hypoxia on Neutrophil Extracellular Traps
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2022-01-034AC
Record Dates: First submitted 2022-08-01; First posted 2022-08-03 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: OSA
Keywords: obstructive sleep apnea; intermittent hypoxia; neutrophil extracellular traps
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleep apnea: 60 moderate-to-severe OSA patients (AHI≧15/hour, 30 obese [BMI>=27] & 30 non-obese [BMI<27])
  Interventions: Other: sleep apnea
- Control: 40 age-, gender-, BMI-matched controls without OSA.

INTERVENTIONS:
Other: sleep apnea — This prospective observational study will enroll 60 moderate-to-severe OSA patients (AHI≧15/hour, 30 obese [BMI>=27] & 30 non-obese [BMI<27]) and 40 age-, gender-, BMI-matched controls without OSA. Venous blood 10 ml will be collected to isolate neutrophils, which are later tested for their ability to produce neutrophil extracellular traps (NETs) under the effect of PMA (phorbol 12-myristate 13-acetate).
  Groups: Sleep apnea

SUMMARY:
This prospective observational study will enroll 60 moderate-to-severe OSA patients (AHI≧15/hour, 30 obese [BMI>=27] & 30 non-obese [BMI<27]) and 40 age-, gender-, BMI-matched controls without OSA. Venous blood 10 ml will be collected to isolate neutrophils, which are later tested for their ability to produce neutrophil extracellular traps (NETs) under the effect of PMA (phorbol 12-myristate 13-acetate). The test will be repeated if OSA patients receive CPAP therapy (continous positive airway pressure therapy).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common disease, affecting around one billion people worldwide. This disorder is characterized by repetitive upper airway collapse during sleep, thereby leading to intermittent hypoxia (IH). The severity of OSA is gauged by AHI(apnea-hypopnea index), which can be determined by a sleep test, polysomnography. Literature revealed OSA confers a higher risk for incident pneumonia and sepsis-related adverse outcomes, suggestive of defective immunity in those patients. CPAP therapy (continous positive airway pressure therapy) is the mainstay treatment for OSA. This research is aimed to investigate the impact of IH on the ability of neutrophils to produce neutrophil extracellular traps (NETs). We will enroll 60 moderate-to-severe OSA patients (AHI≧15/hour, 30 obese [BMI>=27] & 30 non-obese [BMI<27]) and 40 age-, gender-, BMI-matched controls without OSA. Venous blood 10 ml will be collected to isolate neutrophils, which are later tested for their ability to produce NETs under the effect of PMA (phorbol 12-myristate 13-acetate).

ELIGIBILITY:
Inclusion Criteria

* Adults with clinical diagnosis of moderate or severe OSA (AHI >=15/hour)
* Must be willing to participate in this study and sign permit

Exclusion Criteria

* Not willing to participate in this study
* Ever treated with continous positive airway pressure (CPAP) or other therapy for OSA
* Age < 20 years
* Have comorbid disease or condition, which could impact immunity (such as malignancy, chemotherapy, immune disease, diabetes etc)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective observational study will enroll 60 moderate-to-severe OSA patients (AHI≧15/hour, 30 obese [BMI>=27] & 30 non-obese [BMI<27]) and 40 age-, gender-, BMI-matched controls without OSA. Venous blood 10 ml will be collected to isolate neutrophils, which are later tested for their ability to produce neutrophil extracellular traps (NETs) under the effect of PMA (phorbol 12-myristate 13-acetate).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
ability to produce neutrophil extracellular traps (NETs) | 0-90 dyas (if receive therapy)
  Venous blood 10 ml will be collected to isolate neutrophils, which are later tested for their ability to produce neutrophil extracellular traps (NETs) under the effect of PMA (phorbol 12-myristate 13-acetate). The test will be repeated if OSA patients receive CPAP therapy (continous positive airway pressure therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ta Chou, MD & Ph.D, Principal Investigator — Taipei Veterans General Hospital, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided